CLINICAL TRIAL: NCT01534585
Title: Phase Ⅰ/Ⅱ Study of Icotinib Hydrochloride Combined With Intensity-modulated Radiotherapy in Nasopharyngeal Cancer
Brief Title: Safety and Efficacy Study of Icotinib With Intensity-modulated Radiotherapy in Nasopharyngeal Carcinoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Taizhou Hospital (Other)
Responsible Party: Principal Investigator, Haihua Yang, Director of Radiotherapy Dept, Taizhou Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YHH-201201
Record Dates: First submitted 2012-02-13; First posted 2012-02-16 (Estimated); Last update posted 2018-04-17 (Actual); Status verified 2018-04

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: nasopharyngeal carcinoma(NPC); Icotinib; Intensity Modulation Radiation Therapy(IMRT)
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — icotinib; Radiotherapy, Intensity-Modulated; TP protocol; Quality of Life

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Icotinib — Oral Icotinib begins on day 1 and continues until completion of radiotherapy. Phase I:The initial plan is to accrue 6 patients to each dose level (125mg, qd and bid and tid) in each cohort. If one or none of six patients have dose limiting toxicity (DLT), then escalation will proceed. If DLT occurs in two or more patients at a dose level, then escalation will be stopped. The dose level below that at which two of six patients experience a DLT is defined as the maximum-tolerated dose. A minimum of 4 weeks of observation is required after completion of radiation within each Icotinib dose level before accrual to the next level.
  Phase II:According to the maximum tolerated dose, 50 patients will been recruited.
  Other Names: Conmana
Radiation: intensity-modulated radiotherapy — The nasopharyngeal regions and upper neck with IMRT plans will be generated and approved for each patient, whereas the low-neck and supraclavicular regions will be used with a conventional anterior field. A total of 70-76Gy at 2.12-2.3Gy/fraction/d will be given to the GTVnx, the GTVnd will receive 66-70Gy at 2.0-2.12Gy/fraction/d, the CTV1 will receive 60-66Gy at 1.8-2.0Gy/fraction/d, and the CTV2 received 56-60Gy at 1.7-1.8Gy/fraction/d with IMRT. The low-neck and supraclavicular regions will receive 50-60Gy at 2.0Gy/fraction/d with conventional radiotherapy. Target prescription dose and critical structures limit dose are planned according to the RTOG0225 trial.
  Other Names: IMRT
Drug: Paclitaxel and Cisplatin — AC that consisted of two cycles of paclitaxel 135 mg/m2 on day 1 plus cisplatin 30 mg/m2 on days 1-3 will start 4 weeks after the end of CRT.
Other: Quality of life — The EORTC QLQ-C30 and H&N35 of the Chinese version, which is obtained from the Quality of Life Unit, EORTC Data Center in Brussels, Belgium, is available and easily completed by our patients are chosen for this study. Patients will complete the questionnaire before treatment and after treatment and one month after treatment and three months after treatment and one year after treatment.
  Other Names: QoL
Genetic: Epidermal growth factor receptor status — EGFR expression and mutation before treatment.
  Other Names: EGFR

SUMMARY:
Nasopharyngeal carcinoma (NPC) is a prevalent disease in southeast of China. Radiation therapy with or without chemotherapy is a standard therapy for nasopharyngeal cancer. Cytotoxic chemotherapy plays an important role in the curative treatment of advanced NPC. However, concurrent chemoradiotherapy increased significantly local and systemic toxic effects, which may preclude many patients from proceeding with combined therapy. The epidermal growth factor receptor(EGFR) gene is amplified in 40% and EGFR protein is overexpressed in over 80% of NPC. EGFR overexpression is also associated with shorter survival following chemoradiotherapy in locoregionally advanced NPC. And some basic researches have proved that EGFR tyrosine kinase inhibitors(TKIs) could increase the radiosensitivity and reduce the epithelial-mesenchymal transition (EMT) in NPC cell line. Moreover, distant metastases has been the major cause of treatment failure in NPC. Icotinib hydrochloride is a novel oral EGFR TKIs with low mammalian toxicity(made in China). But base on toxic effects of Icotinib, it may increase toxic effects about skin and mucosa in combination therapy with Icotinib and Intensity-modulated Radiotherapy (IMRT). The prospective study will assess the tolerability and efficacy of Icotinib combined with IMRT in patients with NPC. This regimen is of great interest and it has potential to alleviate the adverse effects, improve patient compliance and better therapeutic ratio.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histological proof of squamous carcinoma of the nasopharynx.
2. Patients must have ECOG Performance Status of 0-1.
3. Patients should have adequate bone marrow function defined as an absolute peripheral granulocyte count (AGC) of >/= 1500 cells/mm3, platelet count of >/= 100,000 cells/mm3; adequate hepatic function with bilirubin </= 1.5mg/dl, AST and ALT </= 2x the upper limit of normal; serum creatinine </= 1.5mg/dl, creatinine clearance >/= 50 ml/min and INR 0.8 - 1.2.
4. Patients must sign a study specific informed consent form prior to study entry.

Exclusion Criteria:

1. Evidence of metastases by clinical or radiographic examinations.
2. History of malignancy other than non-melanoma skin cancer.
3. Prior chemotherapy or anticancer biologic therapy for any type of cancer, or prior radiotherapy to the head and neck region except for radioactive iodine therapy.
4. Patients with uncontrolled intercurrent disease.
5. Patients with currently active malignancy.
6. Pregnant or lactating women Female patients of childbearing potential who are unwilling to practice adequate contraception during study treatment and for two months after the last administration of study drug.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2012-02; Primary Completion 2013-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Phase I: the maximum tolerated dose of Icotinib in combination with IMRT for NPC | 30 days
Phase II: 2 years locoregional control rate | Two years

SECONDARY OUTCOMES:
The overall response rate (complete and partial response) | 1 month following treatment and then every 3 months
The acute and late toxicity profile associated with the study regimen | 1 month following treatment and then every 3 months
The duration of control of locoregional disease | 1 month following treatment and then every 3 months
Overall survival, disease-free survival, and distant relapse rates | At time of locoregional disease progression
EGFR status in tissue and blood before treatment | 2 week of pretreatment

CONTACTS AND LOCATIONS:
Overall Officials: Haihua Yang, MD., Study Director — Department of Radiation Oncology, Taizhou Hospital, Wenzhou Medical College.; Wei Hu, MD., Study Chair — Department of Radiation Oncology, Taizhou Hospital, Wenzhou Medical College.; Wei Wang, BS, Principal Investigator — Department of Radiation Oncology, Taizhou Hospital, Wenzhou Medical College.; Chao Zhou, MD., Principal Investigator — Department of Radiation Oncology, Taizhou Hospital, Wenzhou Medical College.
Locations (1):
- Taizhou Hospital, Wenzhou Medical College, Taizhou, Zhejiang, China